CLINICAL TRIAL: NCT06809712
Title: A Prospective Single-arm Trial on Human Leukocyte Antigen (HLA) Mismatched Unrelated Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Human Leukocyte Antigen (HLA) Mismatched Unrelated Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: MIGHT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: He Huang (Other)
Responsible Party: Sponsor-Investigator, He Huang, Professor, Director of the Bone Marrow Transplantation Center, The First Affiliated Hospital, Zhejiang University School of Medicine, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMU-001
Record Dates: First submitted 2024-10-04; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-10

CONDITIONS: Hematologic Disease
Keywords: Hematopoietic cell transplantation; HLA mismatch; Hematologic diseases
MeSH Terms: conditions — Hematologic Diseases | interventions — Busulfan; Cyclophosphamide; fludarabine; fludarabine phosphate; Semustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HLA mismatch (Experimental): Myeloablative conditioning regimen was used when patient is below 50 and with a HCT-CI score <2; Reduced intensity conditioning regimen was used when patient is over 50 or with HCT-CI score ≥2.
  Interventions: Drug: Busulfan (Busulfex); Drug: Cyclophosphamide (CTX); Drug: Fludarabine (Fludara); Drug: Semustine (MeccNU)

INTERVENTIONS:
Drug: Busulfan (Busulfex) — Myeloablative conditioning: Busulfan (Bu，3.2 mg/kg/d IV -8d ~-6d); Reduced intensity conditioning: Busulfan (Bu，3.2 mg/kg/d IV -7d~-5d);
Drug: Cyclophosphamide (CTX) — Myeloablative conditioning: Cyclophosphamide (Cy，1.8g/m2, -5d, -4d) Cyclophosphamide is not used for reduced intensity conditioning
Drug: Fludarabine (Fludara) — Myeloablative conditioning: Fludarabine (Flu，30 mg/m2/d IV -6d ~ -2d); Reduced intensity conditioning: Fludarabine (Flu，30mg/m2 /d IV -10d~-5d);
Drug: Semustine (MeccNU) — For both myeloablative and reduced intensity conditioning:
  Semustine (MeCCNU: 250 mg/m2 orally-3d)

SUMMARY:
This study is a single center, prospective, single arm exploratory clinical trial that includes patients with hematological malignancies who are indicated for allogeneic hematopoietic stem cell transplantation (allo HSCT) but lack suitable donors. This project plans to use highly mismatched unrelated HLA mismatched donors. Ultimately, an unrelated human leukocyte antigen (HLA) mismatched allo HSCT transplantation plan will be established to improve the disease prognosis of this group of patients and truly enter the era of "everyone has a donor" for allo HSCT.

DETAILED DESCRIPTION:
This study is a single center, prospective, single arm exploratory clinical trial that includes patients with hematological malignancies who are indicated for allogeneic hematopoietic stem cell transplantation (allo HSCT) but lack suitable donors. This project plans to use highly mismatched unrelated HLA mismatched donors. Ultimately, an unrelated human leukocyte antigen (HLA) mismatched allo HSCT transplantation plan will be established to improve the disease prognosis of this group of patients and truly enter the era of "everyone has a donor" for allo HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-60 years old) with hematological malignancies and indications for hematopoietic stem cell transplantation;
* Non blood donors without human leukocyte antigen (HLA) high-resolution typing ≥ 9/10, or those who have difficulty finding non blood donors due to urgent medical conditions;
* No suitable HLA matching haploidentical donor available;
* There are suitable unrelated HLA mismatched (HLA high-resolution typing<9/10) donors;
* The subjects or their legal representatives shall sign an informed consent form before the start of the clinical study.

Exclusion Criteria:

* Patients with severe liver and kidney function (alanine aminotransferase>2.5 times the upper limit of normal, blood creatinine>1.5 times the upper limit of normal) and cardiopulmonary dysfunction (New York Heart Association (NYHA) III/IV heart function, ejection fraction<50%, severe obstructive or restrictive ventilation dysfunction);
* Merge active infections;
* Eastern Cooperative Oncology Group Performance Status (ECOG) score ≥ 2 points;
* Secondary tumors with merged activity;
* Severe central nervous system or mental illness leading to the inability to autonomously choose to enter or exit clinical trials;
* Combine other allo hematopoietic stem cell transplantation (HSCT) contraindications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1-year
  Overall survival (OS) after allogeneic hematopoietic cell transplantation is defined as the proportion of patients who are alive at a specified time point following the transplantation, regardless of disease status or cause of death.

SECONDARY OUTCOMES:
Neutrophil engraftment rate | 28-days
  The 28-day neutrophil engraftment rate is assessed, with neutrophil engraftment defined as achievement of an absolute neutrophil count (ANC) of ≥ 0.5 × 10⁹/L for three consecutive days.
Platelet engraftment rate | 28-days
  The 28-day platelet engraftment rate is assessed, with platelet engraftment defined as achievement of a platelet count of ≥ 20 × 10⁹/L without transfusion support for at least seven consecutive days.
GVHD | 180 days and 2 year
  Cumulative incidence of aGvHD and cGvHD in different target organs and overall population.
Relapse | 1-year
  Cumulative incidence of disease relapse after transplantation.
Progression-free survival | 1-year
  Progression-free survival (PFS) after allogeneic hematopoietic cell transplantation is defined as the length of time a patient survives without evidence of disease progression or relapse following the transplantation.
Graft-versus-host disease (GVHD)-free, relapse-free survival (GRFS) | 1-year
  Graft-versus-host disease (GVHD)-free, relapse-free survival (GRFS) after allogeneic hematopoietic cell transplantation is defined as the time a patient survives without experiencing grade III-IV acute GVHD, severe chronic GVHD, relapse, or death.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No